CLINICAL TRIAL: NCT04691440
Title: Hyperbaric Oxygen Treatment in Humans With Gram Positive Cocci Endocarditis"
Brief Title: Hyperbaric Oxygen Treatment in Humans With Gram Positive Cocci Endocarditis
Acronym: ENDOHOT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ole Hyldegaard (Other)
Collaborators: Rigshospitalet, Denmark (Other); Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Ole Hyldegaard, Chief Consultant, MD, Ph.D., Department of HBO, Rigshospitalet, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDOHOT TRIAL - RH; 2019-000857-29 (EudraCT Number)
Record Dates: First submitted 2020-12-18; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Infectious Endocarditis
MeSH Terms: conditions — Endocarditis, Subacute Bacterial | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBOT (Experimental): Hyperbaric oxygen breathing at 2.4 atm.abs for 90 minutes. The course of hyperbaric oxygen treatment comprises a total of 6 pressure exposures, distributed 2 times daily, for 3 days.
  Interventions: Drug: Hyperbaric oxygen

INTERVENTIONS:
Drug: Hyperbaric oxygen — The course of hyperbaric oxygen treatment comprises a total of 6 pressure exposures, distributed 2 times daily, for 3 days.

SUMMARY:
Infectious endocarditis (IE) is defined as an infection anywhere on the endocardium, most often localised to the cardiac valves. It is an infection with an increasing incidence and in Denmark with 6-700 new cases annually. Approximately 45% of the patients must undergo cardiac surgery with replacement of infected cardiac valves by prosthetic valves.

Recently, the formation of biofilms infections has drawn attention with respect to the effects of hyperbaric re-oxygenation of stricken tissues as anaerobic bacterial metabolism with low levels of activity within the biofilm environment, may be responsible for the development of antimicrobial resistance. Polymorphonuclear leukocytes (PMNs) consume available oxygen in the conversion of oxygen to ROS and in the formation of reactive nitrogen species (RNS) by inducible nitric oxide (iNOS) as PMN's are activated by bacteria.

In pre-clinical context the effect of hyperbaric oxygen treatment (HBOT) in re-oxygenating biofilm related infections have been demonstrated in infected lungs with Pseudomonas aeruginosa and staphylococcus aureus endocarditis.

Adjunctive HBOT has never been offered to patients with IE. However, HBOT may be associated with reduced compliance and side effects, such as equalisation problems of ears and sinuses and confinement anxiety, and the treatment is organizational challenging. On this basis the investigators suggest an initial feasibility study as the basis for a later and larger scaled randomized controlled trial of HBOT in patients with IE.

DETAILED DESCRIPTION:
During antibiotic treatments with the indicated antibiotics the susceptible bacteria are subjected to metabolic changes of the Krebs cycles leading to intrabacterial accumulation of toxic hydroxyl oxygen radicals. The intrabacterial toxic reactive oxygen species (ROS) can subsequently react with DNA, lipids or proteins resulting in damages of those bacterial components adding to the killing of the bacteria. A consequence is that bactericidal antibiotics have reduced activity in infectious foci with poor oxygen supply like in abscesses or in biofilm infections as in IE and/or rapid consumption of oxygen due to PMN influx. The bacterial damages may, if killing is not obtained, result in mutations and selection of antibiotic resistant mutants.

However, these discoveries also provide a possibility for improving the antibacterial effect by increasing the oxygen pressure in the infectious focus. This can be obtained by increasing oxygen tension in the tissues by treating the patients with HBOT - and have been shown in vitro and in vivo pre-clinical experiments. Exposing Pseudomonas aeruginosa biofilm models in vitro to HBOT has proved effective by significantly increasing the bactericidal effect of ciprofloxacin.

More important, in an animal (rats) model of left-sided S. aureus IE on the aortic valves, tobramycin killing effect was significantly improved by adding HBOT as adjunctive therapy. Moreover, the rats revealed a reduced inflammatory response and improved clinical scores. No side effects were recorded during that study.

In addition, the HBOT is also believed to improve the antibacterial effect of the PMNs, and thereby add to an enhanced elimination of infectious focus. This is being estimated by measurements of the respiratory burst of the PMNs, as well as their phagocytic capacity right before and right after the HBOT.

ELIGIBILITY:
Inclusion Criteria:

1. Left sided IE with gram positive cocci.
2. IE has been diagnosed according to modified Duke Criteria.
3. Patients must be stable, by means of no need for hemodynamic pressure support.
4. The patient must be able to be seated for the 1.5 hour the HBOT at least two times a day for 3 days.
5. The patient must be able to perform Valsalva's - or Frenzels manoeuvre - to equalize middle ear pressure. As prophylaxis, all patients will receive detumescent nose drops as Otrivin® to facilitate ear- and sinuses equilibration. In the rare event it is still not possible for the patient to equalize pressure, a paracentesis or drainage of the tympanic membrane must be performed by the ear-nose and throat (ENT) doctor. All according to daily practice.
6. The upstart of HBOT must be within the first 2 weeks of relevant antibiotic IE therapy.
7. If a central venous catheter has been inserted, a chest X-ray must confirm no suspicion of pneumothorax.
8. Patients must be >18-years old.

Exclusion Criteria:

1. Claustrophobia that cannot be reversed by mild sedatives.
2. Patients requiring mechanical ventilation.
3. Undrained pneumothorax
4. Pregnancy
5. Unable to follow and understand simple commands
6. Non-compliant

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in baseline characteristics with definite IE. | Up to 12 weeks
  Standard clinical assesments of IE and paraclinical data

CONTACTS AND LOCATIONS:
Overall Officials: Ole Hyldegaard, MD, PHD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark